CLINICAL TRIAL: NCT01984918
Title: Predictors of Colonoscopy Non-attendance and the Efficacy of a Short Message Service (SMS) Reminder to Reduce Non-attendance Rate: A Prospective Randomized Controlled Trial (NAC Study)
Brief Title: Predictors of Colonoscopy Non-attendance and the Efficacy of a SMS Reminder to Reduce Non-attendance Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Aric Josun Hui, Dr., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NAC Study
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Ultilization of Out-patient Colonoscopy Service

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS reminder (Active Comparator): A text message reminder via Short Message Service (SMS) will be sent to remind subjects 7-10 days before his colonoscopy appointment
  Interventions: Other: SMS reminder; Other: Non-SMS reminder
- Non-SMS reminder (No Intervention): No text message reminder via Short Message Service (SMS) will be sent

INTERVENTIONS:
Other: SMS reminder — A text message reminder via Short Message Service (SMS) will be sent to remind subjects 7-10 days before his colonoscopy appointment
  Arms: SMS reminder
Other: Non-SMS reminder — No Stext message reminder via Short Message Service (SMS) will be sent
  Arms: SMS reminder

SUMMARY:
To conduct a prospective randomized controlled study to identify predictors for colonoscopy non-attendance and examine the efficacy of SMS reminder to improve the non-attendance rate.

DETAILED DESCRIPTION:
Implementation of colorectal screening programs has been shown to decrease, the incidence of colorectal cancer due to the early detection and removal of pre-cancerous colonic polyps. Colonoscopy is therefore one of the most common medical procedures performed in the United States with 14 million procedures performed in 2003. Aside from screening, colonoscopy is also essential for other aspects of colorectal cancer management including post-resection surveillance and palliative treatments. Use of computer simulation models showed that the demand for colonoscopy in the United States exceeds current capacity regardless of screening strategy. The incidence of colorectal cancer has been increasing in Hong Kong and has been associated with progressive increase in the colonoscopy waiting times in the public health care system. The progressive increase in the demand for colonoscopy therefore poses a significant burden on the healthcare systems of all developed countries. Methods to increase the capacity and efficiency of the colonoscopy service are needed.

Non-attendance rates of gastrointestinal endoscopy appointments may range from 12% to 27% 5-6 and results in inefficient use of healthcare resources, delay in diagnosis and an increase in waiting times. Adams et al. conducted a prospective cohort study which showed that younger age, long waiting times and referral from a non-gastroenterologist were significantly associated with non-attendance. In an another prospective cohort study, Sola-Vera et al. also showed that the waiting time and source of referral were independent predictive factors for non-attendance 7. Studies on gynecological endoscopy non-attendance revealed that predictors of non-attendance include unemployment, current smokers, younger age, long follow up periods, lower social class, lower education levels and lack of understanding of the endoscopic procedure 8-10.

Telephone reminders have been used to improve non-attendance rates; Adams et al. had decreased the non-attendance rate from 12.2% to 9% after introduction of telephone reminder 1 week prior to the examination. The Mayo clinic open-access endoscopy system, which incorporates a standard telephone reminder 3-7 days prior to the procedure, has a non-attendance rate of only 4.1%.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for an outpatient colonoscopy at the Alice Ho Miu Ling Nethersole Hospital Combined Endoscopy Unit

Exclusion Criteria:

* Age ≤ 18
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2225 (Actual)
Dates: Start 2013-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Non-attendance rate of colonoscopy | Within one year after recruitment
  attendance of colonoscopy on the scheduled colonoscopy date

SECONDARY OUTCOMES:
Predictors of colonoscopy non-attendance | Within one year after recruitment
  different risk factors which may predicts colonoscopy non-attendance
Bowel preparation level | Within one year after recruitment
  bowel preparation level of completed colonoscopy
Predictors of bowel preparation | Within one year after recruitment
  different risk factors which may predicts bowel preparation level

CONTACTS AND LOCATIONS:
Overall Officials: Aric Josun Hui, MD, Principal Investigator — Alice Ho Miu Ling Nethersole Hospital
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong